CLINICAL TRIAL: NCT03257722
Title: A Phase Ib /II Trial of Pembrolizumab and Idelalisib in Patients With Non-small Cell Lung Cancer (NSCLC) Who Have Failed Immune Checkpoint Inhibitor
Brief Title: Pembrolizumab + Idelalisib for Lung Cancer Study
Acronym: PIL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to poor accrual.
Sponsor: Asha Nayak (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Asha Nayak, Professor of Medicine, Augusta University
Organization: Augusta University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCC-16053
Record Dates: First submitted 2017-08-16; First posted 2017-08-22 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Non Small Cell Lung Cancer; Metastasis; Recurrence
Keywords: Non Small Cell Lung Cancer; Metastasis; Recurrence; Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Recurrence | interventions — pembrolizumab; idelalisib

STUDY DESIGN:
Intervention Model Description: This is an open labeled, single arm, interventional study combining standard pembrolizumab (MK-3475, trade name: Keytruda) with investigational agent, idelalisib (trade name: Zydelig) in non-small cell lung cancer (NSCLC). The study will enroll patients in two phases: a dose finding/tolerability assessment phase and an efficacy assessment phase.
  The Phase 1b (modified 3+3 dose escalation) assessment will determine the safe dose of idelalisib in combination with pembrolizumab that down-regulates the activity of T-regulatory function (Treg).
  The Phase 2 efficacy assessment will enroll patients to detect whether idelalisib added to pembrolizumab at the phase 2 recommended dose (P2RD) will result in further objective response.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 Dose Escalation (Experimental): Sequential cohorts of 3 patients will receive pembrolizumab 200 mg intravenously every 3 weeks, in addition to the oral drug, idelalisib, every day for 21 days. The first group of 3 will receive idelalisib 50 mg twice daily; the next cohort will receive idelalisib 100 mg twice daily; the last cohort will receive idelalisib 150 mg twice daily.
  Interventions: Drug: Pembrolizumab; Drug: Idelalisib
- Phase 2 Efficacy (Experimental): All patients in the efficacy assessment phase will be treated with pembrolizumab (200 mg intravenously every 3 weeks) in combination with oral idelalisib (dose not exceeding 150 mg twice daily, per the phase 1 assessment) for 18 weeks before maintenance with pembrolizumab 200 mg intravenously every 3 weeks for up to 2 years, until disease progression or unacceptable toxicity.
  Interventions: Drug: Pembrolizumab; Drug: Idelalisib

INTERVENTIONS:
Drug: Pembrolizumab — Anti PD-1 immunotherapeutic agent, which blocks a protective mechanism on cancer cells to allow the immune system to destroy cancer cells. Administered intravenously (IV).
  Other Names: Keytruda; MK-3475
Drug: Idelalisib — Phosphatidylinositol 3-kinase (PI3K) inhibitor which promotes anti-tumor immune response. Administered orally (PO).
  Other Names: Zydelig; GS-1101

SUMMARY:
This is a phase 1b/2 study to determine the safety and effectiveness of the combination of pembrolizumab and idelalisib in NSCLC patients whose disease has stopped responding to immune therapy. This study is being done to see if adding another immune modulator (idelalisib) to standard pembrolizumab will increase response rates, compared to the response seen with pembrolizumab alone.

DETAILED DESCRIPTION:
This is a phase 1b/2 study to determine the safety and effectiveness of the combination of pembrolizumab and idelalisib in NSCLC patients whose disease has stopped responding to immune therapy. Pembrolizumab is an anti-PD-1 immunotherapy that is given intravenously and is approved for treatment of malignant NSCLC. Idelalisib is the first-in-class oral PI3K-δ inhibitor that is approved for treatment of certain forms of leukemia and lymphoma.

Immune checkpoint inhibitors (such as anti-PD-1) are effective in treating NSCLC as a single agent, but overall response isn't optimal; overall response rates (ORR) are only ~20% on average. The goal of this study is to see whether combining standard therapy with additional immune modulators will increase response rates, compared to the response seen with pembrolizumab monotherapy.

ELIGIBILITY:
All subjects must have documented metastatic or recurrent NSCLC from biopsy. They must have failed or progressed on platinum-based chemotherapy (e.g. cisplatin, carboplatin) as well as immune checkpoint inhibitor therapy (e.g nivolumab or pembrolizumab). Patients with EGFR/ALK mutations/translocations must have failed or progressed on small molecule inhibitor therapies (e.g. erlotinib, afatinib, etc.).

Inclusion Criteria:

* Have at least one measurable lesion
* Have an ECOG Performance Status of 1 or less
* Demonstrate adequate organ function as defined in the protocol.
* Female subjects of childbearing potential must have a negative pregnancy test before starting treatment; they must also be willing to use two methods of birth control or abstain from heterosexual activity for the duration of the study.
* Male subjects must agree to use an adequate method of contraception starting with the first dose of study therapy through the duration of the study.

Exclusion Criteria:

* Is currently receiving study drug in another trial; or has participated in an investigational drug study within 3 weeks of the first dose of treatment.
* Is within 3 weeks of most recent chemotherapy.
* Has a history of hypersensitivity to pembrolizumab or idelalisib, or any of their excipients.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated, stable, brain metastases may participate; carcinomatous meningitis is excluded regardless of clinical stability.
* Has known history of non-infectious pneumonitis that required steroid use or has current pneumonitis.
* Has a known history of active TB (Bacillus Tuberculosis)
* Has active autoimmune disease that has required treatment; known history of Human Immunodeficiency Virus (HIV); known active Hepatitis B or Hepatitis C.
* Has an active infection requiring systemic therapy.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2021-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhonglin Hao, MD, PhD, Principal Investigator — Georgia Cancer Center
Locations (1):
- Georgia Cancer Center at Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Dose Escalation 50mg: Sequential cohorts of 3 patients will receive pembrolizumab 200 mg intravenously every 3 weeks, in addition to the oral drug, idelalisib, every day for 21 days. The first group of 3 will receive idelalisib 50 mg twice daily.
  Only two patients were dosed on this trial at 50mg. Two patients were screen fails.
  Pembrolizumab: Anti PD-1 immunotherapeutic agent, which blocks a protective mechanism on cancer cells to allow the immune system to destroy cancer cells. Administered intravenously (IV).
  Idelalisib: Phosphatidylinositol 3-kinase (PI3K) inhibitor which promotes anti-tumor immune response. Administered orally (PO).
Period: Overall Study
Arm/Group | Phase 1 Dose Escalation 50mg
Started | 2
Completed | 0
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: No patients were enrolled in Phase 2.
Groups:
- Phase 1 Dose Escalation: Sequential cohorts of 3 patients will receive pembrolizumab 200 mg intravenously every 3 weeks, in addition to the oral drug, idelalisib, every day for 21 days. The first group of 3 will receive idelalisib 50 mg twice daily.
  Only two patients were dosed on this trial at 50mg. Two patients were screen fails.
  Pembrolizumab: Anti PD-1 immunotherapeutic agent, which blocks a protective mechanism on cancer cells to allow the immune system to destroy cancer cells. Administered intravenously (IV).
  Idelalisib: Phosphatidylinositol 3-kinase (PI3K) inhibitor which promotes anti-tumor immune response. Administered orally (PO).
Arm/Group | Phase 1 Dose Escalation
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicity (DLT) Events as Assessed by CTCAE v4.03
Description: Modified 3+3 dose escalation design will be used to determine whether the addition of idelalisib to standard pembrolizumab is safe and tolerable in checkpoint inhibitor refractory NSCLC patients. An initial cohort of 3 patients will receive 50 mg twice daily idelalisib with standard pembrolizumab. If none of the 3 patients develop a DLT, another 3 patients will be enrolled. Dose will be escalated or de-escalated based on the occurrence of DLTs. All events will be assessed for possible, probable, or definite relation to idelalisib.
Time Frame: First 9 weeks at each dose level
Population: No patients were enrolled in Phase 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Escalation 50mg
Number analyzed (Participants) | 2
Participants | 2

2. Secondary Outcome: Dose-Finding Assessment for Optimum Dose of Idelalisib in Combination With Pembrolizumab
Description: Determine the phase 2 recommended dose (P2RD) of idelalisib, in combination with pembrolizumab, in patients with checkpoint inhibitor refractory NSCLC. If no more than 1/6 patients in initial cohort develop a DLT, the patients will be tested for T-regulatory cell function suppression (80% suppression in 80% of patients). If dose is escalated or de-escalated, testing will continue to assess for optimal T-reg suppression. The dose at which the tolerability and suppression criteria are both met will be declared the P2RD and the study will proceed to phase 2.
Time Frame: 18-27 weeks
Population: Trial did not progress past Phase 1.
Measure: Number; unit: mg
Arm/Group | Phase 1 Dose Escalation 50mg
Number analyzed (Participants) | 2
mg | NA — Only two participants were dosed at the 50mg dosing level.

3. Secondary Outcome: Overall Response Rates (ORR) to Combination Therapy
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 18 weeks - 2 years
Population: No patients were enrolled in Phase 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Escalation
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Time Frame: Six months
Groups:
- Phase 1 Dose Escalation 50mg: Sequential cohorts of 3 patients will receive pembrolizumab 200 mg intravenously every 3 weeks, in addition to the oral drug, idelalisib, every day for 21 days. The first group of 3 will receive idelalisib 50 mg twice daily.
  Pembrolizumab: Anti PD-1 immunotherapeutic agent, which blocks a protective mechanism on cancer cells to allow the immune system to destroy cancer cells. Administered intravenously (IV).
  Idelalisib: Phosphatidylinositol 3-kinase (PI3K) inhibitor which promotes anti-tumor immune response. Administered orally (PO).
Arm/Group | Phase 1 Dose Escalation 50mg
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT03257722/Prot_SAP_ICF_000.pdf